CLINICAL TRIAL: NCT02426177
Title: Comparison of Oral Labetalol and Oral Nifedipine for Postpartum Hypertension Management
Brief Title: Comparison of Tab.Labetalol and Tab.Nifedipine for Management of Postpartum Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, fariha javed, resident, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DowUHS
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Postnatal Hypertension
Keywords: postpartum hypertension; labetalol in postpartum hypertension; nifedipine in postpartum hypertension
MeSH Terms: interventions — Labetalol; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): tab.labetalol is given to the patient with postpartum hypertension in dose of 100 mg 6 hourly increased to maximum 600 mg in 24 hours
  Interventions: Drug: Labetalol
- group B (Active Comparator): tab.nifedipine is given to the patient with postpartum hypertension in the dose of 10 mg twice a day to maximum dose of 60 mg per 24 hours
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Labetalol — anti-hypertensive agents
  Arms: group A
Drug: Nifedipine — calcium channel blocker ,for lowering blood pressure
  Arms: group B

SUMMARY:
To compare effectiveness of oral labetalol and oral nifedipine for management of postpartum hypertension.

DETAILED DESCRIPTION:
A comparison of oral labetalol and oral nifedipine for management of postpartum hypertension. Which drug is more effective in lowering blood pressures in patient with postpartum hypertension.

ELIGIBILITY:
Inclusion Criteria:

* all women with postpartum hypertension as a continuation of pregnancy induced hypertension,eclampsia, pre-eclampsia or new onset de-novo postpartum hypertension,of any parity.
* age group between 18-48.
* after informed consent.

Exclusion Criteria:

* all women with chronic hypertension, uncontrolled and un treated medical disorders will be excluded.
* conditions in which drugs labetalol and nifedipine is contraindicated.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure less than 140/90 mm of hg | 24 hours
  less than 140/90 mm of hg

CONTACTS AND LOCATIONS:
Overall Officials: fariha javed, mbbs, Principal Investigator — Dow University of Health Sciences